CLINICAL TRIAL: NCT02444637
Title: Open Label Trial of Rivastigmine Patch in Subjects With Mild to Moderate Stage Alzheimer's Disease Having Coexisting Small Vessel Cerebrovascular Disease
Brief Title: Open Label Trial of Rivastigmine Patch in Subjects With Mild to Moderate Stage AD Having Coexisting svCVD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Neuroscience Institute (Other)
Responsible Party: Principal Investigator, Dr Nagaendran Kandiah, Senior Consultant, Department of Neurology, National Neuroscience Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RACE_1.0
Record Dates: First submitted 2015-04-28; First posted 2015-05-14 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Alzheimer Disease; CVA (Cerebrovascular Accident)
MeSH Terms: conditions — Alzheimer Disease; Stroke | interventions — Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rivastigmine (Exelon) Patch (Experimental): For the first 4 weeks of the study, subjects will receive Rivastigmine patch 4.6mg/24 hours. Thereafter, subjects will receive Rivastigmine patch 9.5mg/24 hours.
  Interventions: Drug: Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine
  Other Names: Exelon

SUMMARY:
Rivastigmine, an acetylcholinesterase inhibitor which has been approved by FDA & HSA, is authorized for use in the treatment of mild to moderate dementia of the Alzheimer's type.

In this trial, the investigators will be studying the effectiveness of Rivastigmine in subjects with AD and cerebrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50-85 years
* Diagnosis of dementia of the Alzheimer's type according to the National Institute of Ageing-Alzheimer's Association Criteriah
* MRI brain (with T2 or FLAIR sequences) performed within a 12 month period from time of recruitment demonstrating the presence of WMH of ≥2 on the Fazekas scale (Score range of 0-3 wherein a score of 1 indicates mild WMH, 2 indicates moderate WMH and 3 indicates severe WMH).i
* Clinical Dementia Rating score of 1-2j
* Mini-Mental State Examination (MMSE) scores of 12-26 inclusivek
* English or Mandarin speaking, literate participants

Exclusion Criteria:

* Severe neurological, psychiatric or systemic disease which in the opinion of the clinician could interfere with trial assessments
* The use of any investigational drugs, new psychotropic or dopaminergic agents, cholinesterase inhibitors or anti-cholinergic agents during the 4 weeks prior to recruitment
* Known skin allergy or previous allergic reaction to Rivastigmine patch

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Demonstrated Benefit in Global and Cognitive Measures | 2 Years

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 Years

CONTACTS AND LOCATIONS:
Locations (1):
- National Neuroscience Institute, Singapore, Singapore